CLINICAL TRIAL: NCT01005004
Title: Phase I Study of the Safety and Preliminary Efficacy of Intracerebral Transplantation of HuCNS-SC® Cells for Connatal Pelizaeus-Merzbacher Disease (PMD)
Brief Title: Study of Human Central Nervous System (CNS) Stem Cells Transplantation in Pelizaeus-Merzbacher Disease (PMD) Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CL-N01-PMD
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Pelizaeus-Merzbacher Disease
Keywords: PMD; stem cells; Pelizaeus-Merzbacher Disease; human stem cells; central nervous system stem cells
MeSH Terms: conditions — Pelizaeus-Merzbacher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HuCNS-SC cells (Experimental): Intracerebral implantation of HuCNS-SC via direct injection during surgery
  Interventions: Biological: HuCNS-SC cells

INTERVENTIONS:
Biological: HuCNS-SC cells — intracerebral transplantation
  Other Names: Human central nervous system stem cells

SUMMARY:
The purpose of this study is to determine the safety and preliminary effectiveness of human central nervous system stem cells (HuCNS-SC®) transplantation in patients with Connatal Pelizaeus-Merzbacher Disease (PMD).

DETAILED DESCRIPTION:
Enrolled subjects will be transplanted with HuCNS-SC cells into the brain and will receive immunosuppression for nine months. The study observation period is for one year after transplant surgery. Thereafter, subjects will be enrolled in a long-term observational follow-up study for four years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of connatal PMD
* Molecular genetic confirmation of mutation in the proteolipid protein 1 (PLP1) gene
* MRI consistent with PMD as interpreted by a qualified neuroradiologist

Exclusion Criteria:

* Other significant congenital brain abnormality not related to PMD
* Previous participation in gene transfer or cell transplant trial
* Presence of neurological signs and symptoms not consistent with PMD
* Current or prior malignancy
* Prior organ, tissue or bone marrow transplant

Ages: 6 Months to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety assessment through clinical neurological and MRI evaluation. | one year post transplant

SECONDARY OUTCOMES:
MRI examination for post-transplant myelination | one year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — StemCells, Inc.
Locations (1):
- University of California, San Francisco, San Francisco, California, United States